CLINICAL TRIAL: NCT06590597
Title: Effectiveness of an Educational Intervention to Improve Knowledge, Attitudes and Practices for the Prevention of Malaria in the Embera Katio Population of the Department of Cordoba
Brief Title: Improving Knowledge, Attitudes and Practices for Malaria Prevention in the Embera Katio Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, MARIA DE LOS ANGELES RODRIGUEZ GAZQUEZ, Ph.D in Public Health, Universidad de Antioquia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEI-FE 2021-37
Record Dates: First submitted 2024-05-31; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GRUPO EXPERIMENTAL (Experimental): GROUP RECEIVING EDUCATIONAL INTERVENTION
  Interventions: Behavioral: EDUCATIONAL INTERVENTION FOR MALARIA PREVENTION
- GRUPO CONTROL (No Intervention): GROUP RECEIVING USUAL CARE

INTERVENTIONS:
Behavioral: EDUCATIONAL INTERVENTION FOR MALARIA PREVENTION — The intervention consisted of 4 modules administered in the same number of face-to-face sessions in which educational strategies such as classes, guided discussions, workshops and a booklet designed for the study were used.
  Arms: GRUPO EXPERIMENTAL

SUMMARY:
Objective: To evaluate the effectiveness of an educational intervention compared to regular education in improving knowledge, attitudes and practices (KAP) for the prevention of malaria among indigenous people of the Embera Katío ethnic group in the department of Córdoba (Colombia). Methods: Intervention study with a quasi-experimental design with a control group carried out in three phases: (I) design of the educational intervention, (II) validation of the content of the educational intervention by expert judgement, and (III) implementation of a quasi-experimental study with two groups: intervention (n=60) and control (n=58). The intervention consisted of 4 modules delivered in an equal number of face-to-face sessions using educational strategies such as lectures, guided discussions, workshops, and a primer designed for the study. The control group received the usual education provided by the Ministry of Health. The Pan American Health Organization's instrument "Survey on knowledge, attitudes and practices in addressing malaria in indigenous communities" was used to measure for pre-intervention and post-intervention knowledge, attitudes, practices, and total scores. Results: In the content validation phase by expert jurors, it was found that the four modules obtained adequate content validity indexes ranging between 0.83 and 0.90. The general linear repeated measures models showed a positive effect of the educational intervention on the KAP scores (p<0.001), indicating an effect size of 91% in knowledge, 49% in attitudes, 85% in practices and 93% of the total score. Conclusion: The educational intervention was effective in improving knowledge, attitudes and practices for malaria prevention in the indigenous population of the Embera Katío community in the Department of Córdoba.

DETAILED DESCRIPTION:
From the review of articles about educational interventions to improve KAPs regarding malaria prevention in indigenous communities, an educational intervention was designed that was initially presented to the leaders of the community object of study, who provided their input and knowledge and which were incorporated to the final intervention. This educational intervention was structured into four modules to be administered in an equal number of face-to-face sessions, once per week and lasting three hours per session. The contents addressed per session were: (i) Definition of the disease, its signs and symptoms, (ii) Forms of the infection, (iii) Breeding sites of the vector, and (iv) Preventive actions to reduce the risk of infection. Each module was designed employing educational strategies, such as master classes, guided discussions, workshops, drawings, and use of a printed booklet, designed bearing in mind the observations made by indigenous authorities from the Emberá Katío community, who were consulted to know their perceptions and suggestions about the intervention. Each educational session began with a welcome greeting and assessment of prior knowledge, then the planned theme was developed and, finally, an activity was assigned to be developed at home and socialized during the following session.

ELIGIBILITY:
Inclusion Criteria:

Living in the Alto Sinú region Belonging to the Embera Katio community

Exclusion Criteria:

Failure to attend one of the sessions scheduled to receive the intervention Incomplete response to at least 20% of the questionnaire Voluntary withdrawal from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
IMPROVING KNOWLEDGE, ATTITUDES AND PRACTICES FOR MALARIA PREVENTION | 6 MONTHS
  SCORES ON KNOWLEDGE, ATTITUDES AND PRACTICES

CONTACTS AND LOCATIONS:
Overall Officials: MARIA Rodríguez Gázquez, Study Director — Universidad de Antioquia
Locations (1):
- CORDOBA, Montería, Departamento de Córdoba, Colombia

IPD SHARING:
Plan to Share IPD: No